CLINICAL TRIAL: NCT02914132
Title: Safety and Performance Evaluation of the Seraph® 100 Microbind® Affinity Blood Filter for Reducing Bacteremia in Patients on Hemodialysis
Brief Title: Safety Evaluation of Seraph® 100 to Reduce Bacteremia in Patients on Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ExThera Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP001
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2018-01

CONDITIONS: Bacteremia; Bacterial Infection
MeSH Terms: conditions — Bacteremia; Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Seraph 100 Filter (Other): Renal replacement patient with bacteremia.
  Interventions: Device: Seraph 100 Filter

INTERVENTIONS:
Device: Seraph 100 Filter — Treatment of renal replacement therapy patients with bacteremia.
  Other Names: Seraph 100

SUMMARY:
The purpose of this study is to determine whether the Seraph® 100 Microbind® Affinity Blood Filter (Seraph 100) is safe in the treatment of dialysis patients with bacteremia.

DETAILED DESCRIPTION:
This trial is a prospective, non-randomized study in patients as an adjunctive treatment for blood stream infection (BSI) in patients on renal replacement therapy. The heparin surface being studied is currently marketed on extracorporeal circuits. It has been shown to absorb various types of Gram positive and Gram negative bacteria and to reduce toxins and cytokines in in vitro studies using whole blood. For this study, patients on renal replacement therapy who develop bacteremia will have the Seraph® 100 Microbind® Affinity Blood Filter included in the dialysis circuit for up to 4 hours, on one day, with hourly monitoring. Patients will be followed for 14 days post treatment. Patients will be monitored by vital signs and laboratory indices on the day of treatment and on post procedure day 1, 2, 3, 4, 5, 6, 7 and 14.

ELIGIBILITY:
Inclusion Criteria:

1. Require renal replacement therapy.
2. Be ≥ 18 years old and ≤ 90 years old
3. Positive blood culture and one of the following:

   1. Clinical evidence of a catheter exit site to tunnel infection as evidenced by redness, tenderness or purulence.
   2. Bacteremia is proven with two separate blood cultures from independent vein punctures.
   3. A blood culture with Staphylococcus aureus where the time to positivity is within 14 hours.
   4. Growth from a blood culture taken from the hemodialysis catheter 2 or more hours before the growth of a blood culture drawn peripherally at the same time.

Exclusion Criteria:

1. Have an arteriovenous polytetrafluoroethylene (PTFE) graft.
2. Lack of a commitment to full aggressive support.
3. Have inability to maintain a minimum mean arterial pressure of ≥ 65 mm Hg despite vasopressor therapy and fluid resuscitation.
4. Have had chest compressions as part of cardiopulmonary resuscitation (CPR)
5. Have had an acute myocardial infarction (MI) within the past 3 months.
6. Have had serious injury within 36 hours of screening.
7. Have uncontrolled hemorrhage.
8. Are not expected to live > 14 days.
9. Have malignancy and are not expected to live 42 days.
10. Have neutropenia (absolute neutrophil count <500 cells/µL).
11. Have Child-Pugh Class C cirrhosis.
12. Have New York Heart Association Class IV Heart Failure or an ejection fraction <30%.
13. Have known Antithrombin III deficiency.
14. Have platelet count <30,000/µL.
15. Cannot have intravenous (IV) supplemental iron halted during trial period.
16. Are currently involved in an investigational drug or device trial.
17. Have been previously enrolled in this clinical trial.
18. Next hemodialysis treatment will not take place for at least 24 hours after enrollment.
19. Serious bleedings and clotting disorders, determined by blood transfusion of > 2 units of packed red blood cells, or, An acute (48 h) hemoglobin decline of at least 2 g/dL, transfusion requirement of >4 units over 48h, objective evidence of bleed, documented by physician.
20. Breast feeding and pregnant women
21. Contraindications for heparin sodium for injection are:

    1. Have heparin sensitivity
    2. Severe thrombocytopenia.
    3. With an uncontrolled active bleeding state, except when this is due to disseminated intravascular coagulation
    4. In whom suitable blood coagulation tests, e.g. whole blood clotting time, partial thromboplastin time, etc cannot be performed at appropriate intervals (this contraindication refers to full-dose heparin; there is usually no need to monitor coagulation parameters in patients receiving low-dose heparin)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02; Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan T Kielstein, MD,FASN,FERA, Principal Investigator — Academic Teaching Hospital Braunschweig
Locations (4):
- Germany (4):
  - Klinikum Braunschweig, Braunschweig
  - Universitaetsklinikum-Frankfurt, Frankfurt
  - Medizinische Hochschule-Hannover, Hannover
  - Universitatsklinikum Muenster, Münster

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eden G, Schmidt JJ, Buttner S, Kumpers P, Hafer C, Rovas A, Koch BF, Schmidt BMW, Kielstein JT. Safety and efficacy of the Seraph(R) 100 Microbind(R) Affinity Blood Filter to remove bacteria from the blood stream: results of the first in human study. Crit Care. 2022 Jun 17;26(1):181. doi: 10.1186/s13054-022-04044-7. PMID 35715801

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Seraph 100 Filter
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled in the study
Arm/Group | Seraph 100 Filter
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 15

OUTCOME MEASURES:

1. Primary Outcome: Demonstrate Safety of the ExThera Medical Seraph® 100 Microbind® Affinity Blood Filter in a Hemodialysis Circuit Assessed by Rate of Adverse Events.
Description: Demonstrate safety of the ExThera Medical Seraph® 100 Microbind® Affinity Blood Filter in a hemodialysis circuit assessed by rate of adverse events. No adverse events occured
Time Frame: 14 days
Measure: Number; unit: Percent participants w adverse event
Arm/Group | Seraph 100 Filter
Number analyzed (Participants) | 15
Percent participants w adverse event | 0

2. Secondary Outcome: Reduction of Bacteria in Blood Passed Through the Seraph 100 Filter.
Description: Pathogen reduction of > 40 % as CFU/mL or an increase in time to positivity (TTP) of > 22 minutes in blood passed through the Seraph 100 Filter
Time Frame: 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Seraph 100 Filter
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: 4 hour treatment and 14 day followup
Arm/Group | Seraph 100 Filter
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT02914132/Prot_SAP_000.pdf